CLINICAL TRIAL: NCT03851809
Title: A Randomized Controlled Trial of Wendan Decoction as a Palliative Treatment for Acute Brain Injury
Brief Title: Safety and Efficacy of Wendan Decoction in Acute Moderated to Severe Brain Injury
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Taichung Tzu Chi Hospital (Other)
Responsible Party: Principal Investigator, Borren Huang, Director of Neurosurgery department, Taichung Tzu Chi Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REC103-26
Record Dates: First submitted 2019-02-13; First posted 2019-02-22 (Actual); Last update posted 2019-02-22 (Actual); Status verified 2019-02

CONDITIONS: Acute Brain Injury
Keywords: traditional chinese medicine combination treatment
MeSH Terms: conditions — Brain Injuries

STUDY DESIGN:
Intervention Model Description: randomized clinical trial
Masking Description: no masking design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- neurologic intensive care in acute brain injury (Experimental): With the guidance of Taiwan Neurosurgical Society and Taiwan Neurological Society, patients in the control group were given the consistent treatment. (http://www.neurosurgery.org.tw/nsr/tbi/main.htm and http://www.stroke.org.tw/guideline/guideline_1.asp). The intensive treatments were established according to the traumatic brain injury treatment guidelines and spontaneously intracerebral hemorrhage general treatment principles from these two society in Taiwan.
  Interventions: Drug: Wendan decoction combination in acute brain injury

INTERVENTIONS:
Drug: Wendan decoction combination in acute brain injury — In the intervention group, traditional Chinese medicine was given between 14 days of onset and TCM was used 1 month at least in intervention group.

SUMMARY:
Efficacy and safety of Traditional Chinese Medicine (Wendan decoction) combined with conventional neurologic intensive care in patients with acute moderated to severe brain injury in early stage - A randomized controlled study.

DETAILED DESCRIPTION:
This study adopted a prospective, randomized controlled design. All eligible patients included in the study agreed to participated and signed the informed consent from and the study procedures were approved by the ethical committee of Taichung Tzu Chi general hospital (REC103-26). Patients were recruited from the neurosurgery department of Taichung Tzu Chi general hospital between June 2014 and July 2015. A total of 60 patients were enrolled in this study and randomized into intervention group and control group. All patients of both groups were enrolled within 14 days after episode and a follow-up interview until 6 months from the onset. The intervention group mean regular neuro-intensive care combined TCM and the intervention group mean only neuro-intensive care. But there are 7 patients in intervention group and 12 patients in control group quit out this study

ELIGIBILITY:
Inclusion Criteria:

* traumatic brain injury or spontaneously intracerebral hemorrhage within 14 days of onset;
* an initial score of 3-12 points of GCS score;
* adults between 18 to 80 years old;
* and signed informed consent form.

Exclusion Criteria:

* after 14 days of onset;
* a history of previous TBI or stroke;
* intracranial aneurysm or arteriovenous malformation ruptured;
* combination other major organ injury (heart, lung, intra-abdomen organ, pelvic fracture, major vessels);
* other severe disease such as heart or kidney failure;
* previous diagnosed cancer; and pregnant women.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-06-01 (Actual); Primary Completion 2015-07-31 (Actual); Study Completion 2016-01-31 (Actual)

PRIMARY OUTCOMES:
Ventilator use | 1 month
  how many days of ventilator use
ICU stay | 1 month
  how many days of ICU stay
Glasgow coma scale | 1 month
  from 3 to 15 , higher value indicate better outcome
Disability rating scale | 1 month
  from 0 to 29 , higher value mean worse outcome
modified Rankin scale | 1 month
  from 0 to 6 , 0 mean normal and 6 mean dead , higher value indicated worse outcome
mortality | 1 month
  between 1 month mortality

SECONDARY OUTCOMES:
Glasgow coma scale | 6 month
  from 3 to 15 , higher value indicate better outcome
modified Rankin scale | 6 month
  from 0 to 6 , 0 mean normal and 6 mean dead , higher value indicated worse outcome
Disability rating scale | 6 month
  from 0 to 29 , higher value mean worse outcome
Barthel index | 6 months
  from 0 to 100 , higher value mean independency daily life care and better outcome

IPD SHARING:
Plan to Share IPD: No